CLINICAL TRIAL: NCT06855030
Title: The Effect of Basic Body Awareness Therapy on Posture, Trunk Proprioception, Clinical Parameters of Scoliosis and Body Awareness in Adolescents With Idiopathic Scoliosis
Brief Title: Effects of Body Awareness Therapy on Posture, Trunk Movement, Scoliosis & Body Awareness in Adolescents With Scoliosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gözde Yagci (Gür) (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Sponsor-Investigator, Gözde Yagci (Gür), Prof. Dr., Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HU-SNYaylaci-001
Record Dates: First submitted 2025-02-24; First posted 2025-03-03 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-03

CONDITIONS: Adolescent Idiopathic Scoliosis (AIS)
Keywords: scoliosis; awareness; proprioception; Physiotherapy
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Intervention Model Description: In this study, treatment duration is planned to be 16 weeks. The Scientific Exercises Approach to Scoliosis (SEAS) group will receive 60 minutes of SEAS in the clinic once a week, along with a 40-minute home exercise assignment. The other group will receive 30 minutes of SEAS and 30 minutes of Basic Body Awareness Therapy (BBAT) in the clinic onca a week, and both SEAS and BBAT exercises for 20 minutes each as home assignments.
  Non-drug clinical research and method comparison clinical research.
Who Masked: Participant
Masking Description: Participant's parents.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SEAS group (Experimental): Individuals including this group will only be applied scoliosis specific exercises for treatment. Scientific Exercise Approach to Scoliosis (SEAS) approach will be used. These individuals will be followed in the clinic once a week for 60 minutes. The rest of the week, they will complete their program at home for 40 minutes.
  Interventions: Other: Scoliosis Specific Exercise
- BBAT group (Active Comparator): Individuals in this group will receive Basic Body Awareness Therapy (BBAT) in addition to scoliosis-specific exercises. Individuals in the BBAT group will be seen in the clinic once a week and will receive 30 minutes of BBAT in addition to 30 minutes of SEAS. They will perform their exercises at home for a total of 40 minutes, consisting of 20 minutes of BBAT and 20 minutes of SEAS. Total treatment duration will be the same for each group.
  Interventions: Other: Scoliosis Specific Exercise; Other: Basic Body Awareness Therapy

INTERVENTIONS:
Other: Scoliosis Specific Exercise — In the first session, the individual and their family will learn about AIS, the specific curvature, and the treatment process. They will also be taught correct posture and active self-correction, which means finding the best alignment in three planes. Once the individual becomes confident in their self-correction, they will start exercises. In the SEAS method, exercises begin in a sitting position, and as the individual improves, the exercises will be made more challenging and suited to their level. The rehabilitation protocol includes exercises in standing, squatting, single-leg stance, and on the floor. In each session, previous exercises will be reviewed, and new ones will be added. Individuals will be reminded to practice active self-correction during exercises and daily activities. In literature, there is no fixed protocol for exercise duration and frequency, but it is recommended to do exercises 2-3 times a week for 45 minutes or 20 minutes daily.
  Other Names: SEAS group
Other: Basic Body Awareness Therapy — Body awareness movements will be performed in lying, sitting, and standing positions. Then, they will be varied by incorporating walking, running, and voice use. The patient will be asked to perform these movements with a specific rhythm and coordination. BBAT aims to enhance body awareness and create a more realistic body image by normalizing posture, balance, and muscle tension. The training process will involve gradually increasing awareness of the relationship with the floor, the vertical axis, centering, breathing, and flow. During this therapy process, the goal is to improve the individual's awareness of themselves and their surroundings, helping them adopt the "here and now" experience and later apply it in daily life. At the end of each session, time will be given for the patient to respond to their experience and express their thoughts. There is variability in the application duration in the literature.
  Other Names: BBAT group
  Arms: BBAT group

SUMMARY:
Adolescent idiopathic scoliosis (AIS) is a complex deformity of the spine, and its cause remains unknown. AIS can have negative physical, psychological, and social effects on an individual's health. There are two main treatment options for AIS: surgical and conservative approaches, including observation, exercise, and bracing. Scoliosis-specific exercises (SSE) refer to globally recognized, evidence-based exercise approaches.

In this study, the Scientific Exercise Approach to Scoliosis (SEAS), one of the SSE methods, will be used. SEAS consists of individualized active self-correction exercises combined with functional movements. Additionally, the Basic Body Awareness Therapy (BBAT) method will also be applied. BBAT is a body-focused, comprehensive approach that incorporates slow, rhythmic movements and breath control.

Both groups will attend supervised sessions in the clinic once a week, and home exercises will be assigned for the remaining days. Participants in the SEAS group will receive only SEAS treatment, while those in the BBAT group will receive both SEAS and additional BBAT exercises.

The goal of this clinical study is to investigate the effects of BBAT in addition to a rehabilitation program including SSE, on posture, spatial orientation, trunk proprioception, scoliosis-specific parameters, quality of life, and body in adolescents with IS aged between 10 and 17 years.

The research hypotheses for this study are as follows:

H1: Basic Body Awareness Therapy has an effect on posture in adolescents with idiopathic scoliosis.

H2: Basic Body Awareness Therapy has an effect on spatial orientation in adolescents with idiopathic scoliosis.

H3: Basic Body Awareness Therapy has an effect on trunk proprioception in adolescents with idiopathic scoliosis.

H4: Basic Body Awareness Therapy has an effect on scoliosis-specific clinical parameters in adolescents with idiopathic scoliosis.

H5: Basic Body Awareness Therapy has an effect on both general and scoliosis-specific quality of life in adolescents with idiopathic scoliosis.

H6: Basic Body Awareness Therapy has an effect on body awareness in adolescents with idiopathic scoliosis.

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis (AIS) is a 3-dimensional complex deformity of the spine, involving lateral curvature, axial rotation, and altered sagittal physiological curves, that occurs in children between the ages of 10 and skeletal maturity. AIS is the most common type, accounting for 84-89% of all types of scoliosis. Although there are many studies in the literature on its aetiopathogenesis, the cause is still unknown. AIS causes chronic back pain, muscle imbalance in the trunk, limited spinal movement, weakening of the para spinal muscles, reduced respiratory capacity, and dissatisfaction with physical appearance due to distorted body image.The main concern about scoliosis is progression of the deformity. In the absence of treatment, scoliosis can lead to negative physical, psychological, and social effects on an individual's health Individuals with idiopathic scoliosis (IS) are known to have a lower quality of life than their healthy peers. The progressive nature of the disease can be considered a factor contributing to the decline in quality of life.

There are two main treatment options for IS: surgical and conservative (observation, exercise, brace) approaches. Because of its complex underlying mechanism, IS requires a comprehensive conservative treatment approach. The current preventive approach to scoliosis rehabilitation is scoliosis-specific exercises (SSE). SSE is the general term for globally recognized evidence-based exercise approaches. In this study, the Scientific Exercise Approach to Scoliosis (SEAS), a school of thought focused on active self-correction, will be used. SEAS is an exercise program designed to enhance spinal stability through individualized, active self-correction without external assistance, integrated into functional exercises.

The three-dimensional deformities in scoliosis lead to musculoskeletal problems such as postural changes, muscle imbalance, sensory disturbances, and deficits in balance and postural stability. As a result, postural control and trunk alignment awareness are impaired. Another factor affecting postural control, vertical perception, is also known to be disrupted in individuals with AIS however, no specific exercise model focuses on this issue.

Basic Body Awareness Therapy (BBAT) is a comprehensive approach that considers the physical, physiological, psychological, and existential aspects of human existence. It includes fundamental functions such as postural stability, relaxed breathing, and awareness. The therapy consists of daily movements like lying, sitting, standing, and walking, aiming to enhance body awareness and develop a more realistic body image by normalizing posture, balance, and muscle tension. The learning process involves gradually increasing awareness of grounding, the vertical axis, breathing, flow, and centering. Individuals are encouraged to focus not only on their movements but also on their experiences while performing them, fostering both physical and mental self-awareness. The slow movements in BBAT integrate postural alignment awareness with breathing, aiming to improve body awareness, movement quality, posture, coordination, balance, postural control, and physical-social functions. It is recommended in the literature that adding BBAT exercises to the rehabilitation program of individuals with AIS may help improve internal body orientation. BBAT's slow and rhythmic movements, which are focused on postural alignment and postural awareness, can help improve the postural control deficits commonly seen in AIS, by improving trunk alignment and proprioception.

The study will include voluntary participants with IS aged between 10 and 17. The individuals will be evaluated twice: at the beginning and at the end of the treatment.

The Cobb angle is the gold standard method for measuring the curve angle on frontal X-ray. Another indicator of scoliosis, trunk rotation, was measured using the forward bending test with a scoliometer. The scoliometer is designed to measure trunk asymmetry and axial trunk rotation. These two values give us the severity of the deformity. Concerns about aesthetic appearance in adolescents with IS lead to a decrease in quality of life and are a primary reason for seeking healthcare. Therefore, we will use the Spinal Appearance Questionnaire (SAQ) for assessing cosmetic appearance. With this questionnaire, we will evaluate the perception of the deformity by the individual, parent and physiotherapist. Posterior Trunk Symmetry Index (POTSI) and Anterior Trunk Symmetry Index (ATSI) are assessment methods used in the coronal plane that can be applied to all age groups and provide an objective measure of the effectiveness of the treatment on postural and body symmetry. For this purpose, we will take front and back photographs of the individual and make measurements based on ATSI and POTSI. It is accepted that increasing proprioceptive capacity can prevent the deterioration of proper posture and the progression of deformity, which is why it is important in individuals with AIS. The Joint Repositioning Test (JRPT) will be used to assess trunk proprioception. Literature reports that the most sensitive angles for assessment in this group are 15° and 30°, so trunk flexion will be measured at these angles. The Neutral Lumbar Positioning Test (LNP) will be used to assess the difficulty individuals experience in repositioning their spines. Spatial orientation was assessed using the Fukuda Stepping Test, which also evaluates dynamic balance. Two questionnaires will be used to assess individuals' body awareness. The first is the Body Awareness Questionnaire (VFA), which explores body responses, individuals' predictions about body processes, the disease process, and the sleep-wake cycle. The second is The Awareness Body Chart (ABC), which evaluates the level of perception and awareness regarding different body parts. The Japanese Scoliosis Questionnaire-27 (SJ-27) was used for scoliosis-related quality of life assessment, and the Pediatric Quality of Life Inventory (PedsQL) was used for general quality of life evaluation.

This study will include two groups. Both groups are required to perform their exercises individually with a physiotherapist in the clinic once a week and continue with a home exercise program on the remaining days of the week. Individuals in the SEAS group will receive 60 minutes of SEAS once a week in the clinic, while the BBAT group underwent the same SEAS program along with an additional 30-minute BBAT session, totaling 60 minutes per session for 16 weeks. Participants in the SEAS group will perform 40 minutes of SEAS exercises at home, while those in the BBAT group will practice 20 minutes of SEAS and 20 minutes of BBAT exercises.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with adolescent idiopathic scoliosis
* Being between the ages of 10 and 17
* Having scoliosis of 15° or greater
* Not having received previous treatment for scoliosis and not receiving any other treatment during this study
* Risser stage 0-4
* Willing to participate in the study

Exclusion Criteria:

* Having any spinal/bone deformity in addition to scoliosis (such as hyperkyphosis, pectus, etc.)
* Wearing a brace
* Having congenital scoliosis
* Having any rheumatological, neuromuscular, neurological, cardiovascular, or pulmonary pathology
* Having a regular history or habit of physical activity
* Having undergone scoliosis surgery

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Trunk Proprioception | 16 weeks
  To evaluate trunk proprioception, three tests will be used. Measurements will be repeated three times for each test, and the average value will be calculated. The obtained angle will be recorded in degrees and referred to as the error angle.
Posture ( perception of deformity severity) | 16 weeks
  For posture assessment, the Spinal Appearance Questionnaire will be used first. It will be completed by the participant, their parent, and the physiotherapist. In this way, the perception of deformity severity will be measured. It is a valid measure for assessing self-image in adolescents with idiopathic scoliosis. This questionnaire includes 11 standardized drawings that represent different severity levels of spinal deformity perception. Additionally, it consists of 22 Likert-scale questions reflecting the patient's impressions and expectations regarding their appearance. Patients select one of five response options for each drawing, with 1 indicating the best and 5 indicating the worst perception. The total score is the sum of all responses, and a higher score indicates a more severe deformity.
Postural Symmetry for Anterior Trunk | 16 weeks
  Anterior Trunk Symmetry Index (ATSI) is another objective method used to assess postural asymmetry in the anterior trunk. Similar to POTSI, ATSI calculations are based on photographs taken in the optimal standing posture. Although reference values for ATSI are available for different age groups, a definitive normal value has not been established. Higher ATSI values indicate increased asymmetry.
Postural Symmetry for Posterior Trunk | 16 weeks
  Posterior Trunk Symmetry Index (POTSI) is an objective and comprehensive method used to evaluate an individual's postural asymmetry. For the calculation of POTSI, photographs will be taken in the optimal standing posture for assessment. The ideal value of the POTSI index is 0, indicating that the trunk is symmetric, while values above 0 represent asymmetry.
Scoliosis-specific parameters | 16 weeks
  For the assessment of scoliosis parameters, curve severity and trunk rotation will be measured. The Cobb angle method, considered the gold standard, will be used to assess the severity of the curve, measured from the individual's antero-posterior X-ray image. The Cobb angle is defined as the angle between the superior endplate of the uppermost vertebra and the inferior endplate of the lowermost vertebra involved in the curve in the coronal plane. A Cobb angle greater than 10° is required for a diagnosis of AIS. The scoliometer will be use to assess axial trunk rotation. It is a type of inclinometer that measures the symmetry of both sides of the trunk and records it in degrees. The value of 0 observed on the scoliometer indicates that the trunk is symmetric, while values above 0 indicate asymmetry. A 5° threshold on the scoliometer is considered significant, with values above it being regarded as meaningful.
Spatial Orientation | 16 weeks
  The Fukuda stepping test will be used to assess spatial orientation. Measurements will be taken between the marked points at the start and end of the test, with displacement distance recorded in centimeters and displacement angle in degrees. A decrease in angle or distance will be considered an improvement. Although there are no reference values for individuals with AIS, it has been emphasized in the literature that this test is effective in demonstrating proprioceptive deficits in this group. This test will provide information about individuals' dynamic proprioception.
Body awareness (Awareness of body responses) | 16 weeks
  The Body Awareness Questionnaire (BAQ) is used to assess individuals' body awareness by exploring body responses, predictions about bodily processes, the disease process, and the sleep-wake cycle. It consists of 18 items and 4 subgroups in a Likert scale format. Participants rate statements from 1 (Not true for me) to 7 (Completely true for me). The total score is calculated by summing the ratings, and an increase in the score indicates improved body awareness.
Body awareness and perception | 16 weeks
  The Awareness Body Chart (ABC) is another tool used to assess body awareness. It includes simple front and back drawings of male and female bodies, divided into 51 regions and 14 body parts. Participants are asked to color these body parts according to awareness levels represented by specific colors. The total score is calculated by summing the points corresponding to the colors, and an increase in the score indicates an improvement in awareness.

SECONDARY OUTCOMES:
Quality of life related to scoliosis | 16 weeks
  In this study, the Japanese Scoliosis Questionnaire-27 (SJ-27) will be used to assess the quality of life specific to scoliosis in individuals. This questionnaire evaluates the quality of life in patients with Adolescent Idiopathic Scoliosis from a broad perspective, including pain and psychosocial issues. Consisting of 27 items, the questionnaire is scored on a scale from 0 (none) to 4 (severe/very high). To calculate the total score, the answers are summed up, with a higher score indicating a lower quality of life. The minimum score a participant can obtain from this questionnaire is 0, and the maximum score is 108. It includes five areas: pain, discomfort while dressing, appearance-related discomfort, anxiety, and difficulty participating in activities. There are 4 questions related to back pain, 7 questions on discomfort while dressing, 4 on physical activity, 6 on self-consciousness, and 6 questions addressing psychological issues such as depression.
General quality of life | 16 weeks
  The Pediatric Quality of Life Inventory (PedsQL) will be administered to both the child and the parent to assess general quality of life. PedsQL is an assessment questionnaire that measures the impact of both the disease and treatment on the individual's physical, psychological, and social functioning, as well as the effect of disease- and treatment-specific symptoms on quality of life. Scales are available for various age ranges. Two forms are required for the individuals in this study, based on their age. Two different parallel versions will be used for children aged 8-12 years and 13-18 years. Both forms have the same content, but the wording in the 8-12 years form is simplified for this age group. The child form, written in the third-person language, will also be filled out by the parent. It consists of 3 domains and 23 items. As the total PedsQL score increases, so does the quality of life. As the total PedsQL score increases, the quality of life improves.
Evaluation of treatment compliance | 16 weeks
  Adherence to home exercise programs during the 16-week treatment period will be evaluated on a scale from 0 to 100. At the end of the treatment, the patient's adherence to exercises will be assessed for both groups with the question, 'During the 16 weeks, what percentage of your daily home exercises did you follow?' and the responses will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Gözde Yağcı, Prof. Dr., Study Director — Hacettepe University; Sena Yaylacı, MSc, PT, Principal Investigator — Hacettepe University
Locations (2):
- Turkey (Türkiye) (2):
  - Faculty of Physiotherapy and Rehabilitation, Hacettepe, Ankara, 06000, Ankara
  - Hacettepe University Faculty of Physical Therapy and Rehabilitation, Orthotics and Biomechanics Clinic, Ankara

IPD SHARING:
Plan to Share IPD: No